CLINICAL TRIAL: NCT06492733
Title: A Pivotal, Single-arm, Multi-centre, Prospective Clinical Investigation to Assess the Efficacy and Safety of the FastWire REvascularisation of Extremities, (For LOWer Limbs) (FREEFLOW).
Brief Title: FastWire REvascularisation of Extremities, (For LOWer Limbs) - FREEFLOW
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Versono Medical Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP002FREEFLOW PIVOTAL
Record Dates: First submitted 2024-07-01; First posted 2024-07-09 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Chronic Total Occlusion of Artery of the Extremities
Keywords: Chronic Total Occlusion; Peripheral; CTO; FastWire System; FastWire wire; intra-luminal; Active wire; Procedure; Device; peripheral vascular disease; critical limb ischemia; CLI; CLTI; critical limb threatening ischemia
MeSH Terms: conditions — Peripheral Vascular Diseases; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- FastWire System - Peripheral (Experimental): This study is to assess the safety and efficacy of the FastWire System. It is intended to assess that the FastWire System can facilitate the intra-luminal placement of conventional guidewires or treatment devices beyond peripheral artery chronic total occlusions (CTOs).
  Interventions: Device: FastWire System - Peripheral

INTERVENTIONS:
Device: FastWire System - Peripheral — The Investigator can use the FastWire System during the procedure to cross CTO Caps and/or to cross multiple lesions.

SUMMARY:
This study is to assess the safety and efficacy of the FastWire System. It is intended to assess that the FastWire System can facilitate the intra-luminal placement of conventional guidewires or treatment devices beyond peripheral artery chronic total occlusions (CTOs)

DETAILED DESCRIPTION:
Single-arm, multi-center, pivotal study to assess the efficacy and safety of the FastWire System in patients who have a chronic total occlusion in their peripheral vasculature causing an ischemic limb. The enrollment will consist of up to 65 patients meeting the inclusion/exclusion criteria.

ELIGIBILITY:
General Inclusion Criteria: Subjects who meet all the following criteria are eligible for this clinical investigation:

1. The patient signed and dated an Informed Consent Form.
2. Aged between 18 years and 85 years (inclusive).
3. Severe claudication assessed as Rutherford category 3 or CLTI assessed as Rutherford category 4 or 5 LEAD.

Angiographic Inclusion Criteria

Unless otherwise specified, the Investigator performing the procedure bases angiographic inclusion on the visual determination of qualification imaging taken at the time of the procedure. Subject must meet ALL the following angiographic inclusion criteria:

1. Angiographic confirmation at the time of the procedure of a de novo CTO below the origin of the superficial femoral artery (SFA) including above the knee or below the knee. (Note: Multilevel CTOs are included as long as the total length from the beginning of the most proximal total occlusion to the end of the most distal total occlusion is less than 40 cm.)
2. 100% stenosis by a visual estimate of angiography at the time of procedure.
3. For below-the-knee CTOs, the target limb shall have at least one patent (<50% stenosis) run-off vessel confirmed by angiography or magnetic resonance angiography at the time of the procedure.

Exclusion Criteria:

Subjects who meet any of the following criteria are not eligible for this clinical investigation:

1. Life expectancy of less than 12 months.
2. Females who are pregnant or lactating (urine test for women of childbearing age).
3. Myocardial infarction or stroke in two months prior to the index procedure.
4. Known, unstable coronary artery disease or other, uncontrolled comorbidity.
5. Any known haemorrhagic or coagulation deficiency.
6. Known sensitivity to nickel, titanium, or their alloys.
7. Evidence of active infection, including but not limited to the target limb.
8. Current use of cocaine or other substances of abuse.
9. Patients who have received any thrombolytic therapy in the last two weeks.
10. History of severe allergy or contraindication, to contrast medium or other medications used during or after endovascular therapy.
11. Subject participating in another study involving an investigational drug or device.
12. Patient has surgery or vascular intervention planned within 30 days of the index procedure.
13. Patient has had a previous peripheral bypass that includes the target vessel.
14. Patient has had a previous intervention in the target CTO (angioplasty, stenting) including previous attempt at time of index procedure.
15. Patient tests positive for coronavirus disease (COVID-2019), as per site standard practice.
16. Estimated Glomerular Filtration Rate (eGFR) of less than 30 ml/min or creatine level >2.5mg/ml.
17. Platelet count < 50,000/μL.

Angiographic Exclusion Criteria

Unless otherwise specified, the Investigator performing the procedure bases angiographic exclusion on a visual determination of qualification imaging taken at the time of the procedure. Subject is excluded if ANY of the following angiographic exclusion criteria is met:

1. For below-the-knee CTOs, a target limb without at least one patent (<50% stenosis) run-off vessel confirmed by angiography or magnetic resonance angiography at the time of the procedure.
2. Has an acute or sub-acute intraluminal thrombus within the target vessel.
3. Aneurysm distal to puncture access site at least twice the reference vessel diameter, located in the index vessel, abdominal aorta, iliac, or popliteal.
4. Has perforation, dissection, or other injury of the access site or index vessel requiring stenting or surgical intervention prior to attempting crossing of the target lesion with the FastWire System.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2024-11-05 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Clinical success (On Day of Procedure) | Day 1
  Ability to facilitate treatment of the target lesion using the FastWire as a crossing device only and by allowing additional devices to cross the CTO as required. This will be angiographically confirmed.
Freedom from Serious Adverse Events | Up to Day 30
  Freedom from Serious Adverse Events related to the use of the FastWire System, at 30 days post procedure:
  * Cardiovascular deaths.
  * Vessel dissection (Grade C or greater) requiring an intervention to resolve.
  * Unplanned index limb amputation.
  * Symptomatic distal embolization is defined as clinical signs or symptoms of distal emboli detected in the treated limb distal to the treated lesion after the index procedure or noted angiographically after the index procedure and requiring mechanical or pharmacologic means to improve flow.

SECONDARY OUTCOMES:
Technical success (On Day of Procedure) | Day 1
  Ability of the FastWire System to be successfully delivered to, cross through, and retrieved from angiographically confirmed chronic total occlusions.
SADE (Up to Day 30) | Up to Day 30
  Freedom from Serious Adverse Device Effects (SADE).
Vessel dissection or bleeding (Within 24 Hours, Max 36 hrs) | Within 24 Hours, Max 36 hrs
  Freedom from Vessel dissection (Grade C or greater) or bleeding within 24 hours (maximum 36 hours) of the index procedure.
Traverse the CTO (On Day of Procedure) | Day 1
  Ability of the FastWire wire to fully traverse the CTO with entry into the distal true lumen without the need for additional guidewires and/or re-entry devices.
Procedural success (On Day of Procedure) | Day 1
  Procedural success, defined as achievement of technical success together with post-procedural patency. Post-procedural patency is defined as less than or equal to 50% residual percent diameter stenosis assessed by visual estimate at the end of the revascularization procedure.
Procedure-related mortality (Up to Day 7 & Day 30) | Up to Day 7 & Day 30
  All procedure related mortality at day 7 post procedure, and all-cause mortality at 30 days post procedure.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - EndoVascular Consultants, Wilmington, Delaware
  - Vascular & Embolization Specialists, Cocoa, Florida
  - Vascular Institute of the Midwest, Davenport, Iowa
  - Cardiovascular Institute of the South-ASC, Gray, Louisiana
  - Dearborn Cardiology, Dearborn, Michigan
  - Vascular Institute of Chattanooga, Chattanooga, Tennessee

IPD SHARING:
Plan to Share IPD: No